CLINICAL TRIAL: NCT01711359
Title: A Randomized, Double-Blind, Active-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib (LY3009104) in Patients With Moderately to Severely Active Rheumatoid Arthritis Who Have Had Limited or No Treatment With Disease-Modifying Antirheumatic Drugs
Brief Title: A Study in Participants With Moderate to Severe Rheumatoid Arthritis
Acronym: RA-BEGIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14062; I4V-MC-JADZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baricitinib + MTX (Experimental): Baricitinib 4 milligram (mg) administered orally once daily through Week 52. Participants received methotrexate (MTX) orally once weekly with dose ranging from 10 to 20 mg per week through Week 52. Starting at Week 24, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily and MTX orally once weekly.
  Interventions: Drug: Baricitinib; Drug: Methotrexate; Drug: Folic Acid
- Baricitinib (Experimental): Baricitinib 4 mg administered orally once daily through Week 52. Participants received MTX placebo orally once weekly through Week 52. Starting at Week 24, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily and MTX orally once weekly.
  Interventions: Drug: Baricitinib; Drug: MTX Placebo; Drug: Folic Acid
- MTX (Active Comparator): MTX administered orally once weekly with dose ranging from 10 to 20 mg per week through Week 52. Participants also received baricitinib placebo orally once daily. Starting at Week 24, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily and MTX orally once weekly.
  Interventions: Drug: Methotrexate; Drug: Baricitinib Placebo; Drug: Folic Acid

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib; Baricitinib + MTX
Drug: Methotrexate — Administered orally
  Arms: Baricitinib + MTX; MTX
Drug: Baricitinib Placebo — Baricitinib placebo administered orally once daily.
  Arms: MTX
Drug: MTX Placebo — MTX placebo administered orally once weekly.
  Arms: Baricitinib
Drug: Folic Acid — Administered orally every day

SUMMARY:
The purpose of this study is to determine whether baricitinib therapy alone is noninferior to methotrexate (MTX) therapy alone in the treatment of moderate to severe active rheumatoid arthritis (RA) in those who have had limited or no treatment with MTX and are naive to other conventional or biologic disease-modifying antirheumatic drugs (DMARDs).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset rheumatoid arthritis (RA) as defined by American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) 2010 Criteria for the Classification of RA
* Have documented history of positive rheumatoid factor and/or cyclic citrullinated peptide (CCP) antibody test
* Have moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints
* Have a C-reactive protein (CRP) or high-sensitivity C-reactive protein (hsCRP) measurement ≥1.2 times the upper limit of normal (ULN)
* Have had limited or no treatment with methotrexate (MTX)

Exclusion Criteria:

* Have received conventional disease-modifying antirheumatic drugs (DMARDs) other than MTX (eg, gold salts, cyclosporine, leflunomide, azathioprine, hydroxychloroquine, sulfasalazine or any other immunosuppressives)
* Are currently receiving corticosteroids at doses >10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization
* Have started treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of study entry or within 6 weeks of planned randomization
* Have started a new physiotherapy treatment for RA in the 2 weeks prior to study entry
* Have ever received any biologic DMARD
* Have received interferon therapy within 4 weeks prior to study entry or are anticipated to require interferon therapy during the study
* Have received any parenteral corticosteroid administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require a parenteral injection of corticosteroids during the study
* Have had 3 or more joints injected with intraarticular corticosteroids or hyaluronic acid within 2 weeks prior to study entry or within 6 weeks prior to planned randomization
* Have active fibromyalgia that, in the investigator's opinion, would make it difficult to appropriately assess RA activity for the purposes of this study
* Have a diagnosis of any systemic inflammatory condition other than RA, such as, but not limited to, juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, active vasculitis, or gout (Participants with secondary Sjogren's syndrome are not excluded.)
* Have a diagnosis of Felty's syndrome
* Have had any major surgery within 8 weeks of study entry or will require major surgery during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the participant
* Have experienced any of the following within 12 weeks of study entry: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking investigational product or could interfere with the interpretation of data
* Are largely or wholly incapacitated permitting little or no self care, such as, being bedridden or confined to a wheelchair
* Have an estimated Glomerular Filtration Rate (eGFR) based on the most recent available serum creatinine using the Modification of Diet in Renal Disease (MDRD) method of <40 milliliter per minute per 1.73 m^2 (mL/min/1.73 m^2)
* Have a history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the ULN or the most recent available total bilirubin ≥1.5 times the ULN
* Have a history of, lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for <5 years
* Have been exposed to a live vaccine within 12 weeks prior to planned randomization or are expected to need/receive a live vaccine during the course of the study (with the exception of herpes zoster vaccination)
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection
* Have had symptomatic herpes zoster infection within 12 weeks prior to study entry
* Have a history of disseminated/complicated herpes zoster (eg, multidermatomal involvement, ophthalmic zoster, central nervous system involvement, postherpetic neuralgia)
* Are immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study
* Have a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Have screening laboratory test values, including thyroid-stimulating hormone (TSH), outside the reference range for the population or investigative site that, in the opinion of the investigator, pose an unacceptable risk for the participant's participation in the study
* Have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator or the sponsor, are clinically significant and indicate an unacceptable risk for the participant's participation in the study
* Have symptomatic herpes simplex at the time of study enrollment
* Have evidence of active or latent tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (153):
- United States (47):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Cajon, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Desert, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boulder, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lewes, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boynton Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Naples, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venice, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vernon Hills, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cumberland, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freehold, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hartsdale, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duncansville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wyomissing, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grapevine, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nassau Bay, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesapeake, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kennewick, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clarksburg, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Franklin, Wisconsin
- Argentina (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quilmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Fernando
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- Belgium (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mons
- Brazil (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goiânia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Canada (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Victoria, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Catherines, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trois-Rivières, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saskatoon, Saskatchewan
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Nauheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayreuth
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gommern
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
- India (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahmedabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Attavar, Mangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belagavi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaipur
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kolkata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lucknow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Delhi
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valeggio sul Mincio
- Japan (23):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Japan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mie
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okinawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Potosí City
- Portugal (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lisbon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto
- Puerto Rico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Germán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ryazan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulyanovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yaroslavl
- South Africa (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloemfontein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenacres
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Somerset West
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stellenbosch
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Sweden (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huddinge
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malmo
- United Kingdom (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cambridge, Cambridgeshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Basingstoke, Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southampton, Hants
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Shields, Tyneside

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Landewe R, Sun L, Chen YF, Daojun M, van der Heijde D. Robust analyses for radiographic progression in rheumatoid arthritis. RMD Open. 2023 Apr;9(2):e002543. doi: 10.1136/rmdopen-2022-002543. PMID 37015757
- [Derived] Taylor PC, Alten R, Alvaro Gracia JM, Kaneko Y, Walls C, Quebe A, Jia B, Bello N, Terres JR, Fleischmann R. Achieving pain control in early rheumatoid arthritis with baricitinib monotherapy or in combination with methotrexate versus methotrexate monotherapy. RMD Open. 2022 Mar;8(1):e001994. doi: 10.1136/rmdopen-2021-001994. PMID 35264432
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] van der Heijde D, Kartman CE, Xie L, Beattie S, Schlichting D, Mo D, Durez P, Tanaka Y, Fleischmann R. Radiographic Progression of Structural Joint Damage Over 5 Years of Baricitinib Treatment in Patients With Rheumatoid Arthritis: Results From RA-BEYOND. J Rheumatol. 2022 Feb;49(2):133-141. doi: 10.3899/jrheum.210346. Epub 2021 Sep 15. PMID 34526397
- [Derived] Emery P, Tanaka Y, Cardillo T, Schlichting D, Rooney T, Beattie S, Helt C, Smolen JS. Temporary interruption of baricitinib: characterization of interruptions and effect on clinical outcomes in patients with rheumatoid arthritis. Arthritis Res Ther. 2020 May 15;22(1):115. doi: 10.1186/s13075-020-02199-8. PMID 32414425
- [Derived] Fleischmann R, Takeuchi T, Schiff M, Schlichting D, Xie L, Issa M, Stoykov I, Lisse J, Martinez-Osuna P, Rooney T, Zerbini CAF. Efficacy and Safety of Long-Term Baricitinib With and Without Methotrexate for the Treatment of Rheumatoid Arthritis: Experience With Baricitinib Monotherapy Continuation or After Switching From Methotrexate Monotherapy or Baricitinib Plus Methotrexate. Arthritis Care Res (Hoboken). 2020 Aug;72(8):1112-1121. doi: 10.1002/acr.24007. PMID 31233281
- [Derived] Smolen JS, Genovese MC, Takeuchi T, Hyslop DL, Macias WL, Rooney T, Chen L, Dickson CL, Riddle Camp J, Cardillo TE, Ishii T, Winthrop KL. Safety Profile of Baricitinib in Patients with Active Rheumatoid Arthritis with over 2 Years Median Time in Treatment. J Rheumatol. 2019 Jan;46(1):7-18. doi: 10.3899/jrheum.171361. Epub 2018 Sep 15. PMID 30219772
- [Derived] Taylor PC, Kremer JM, Emery P, Zuckerman SH, Ruotolo G, Zhong J, Chen L, Witt S, Saifan C, Kurzawa M, Otvos JD, Connelly MA, Macias WL, Schlichting DE, Rooney TP, de Bono S, McInnes IB. Lipid profile and effect of statin treatment in pooled phase II and phase III baricitinib studies. Ann Rheum Dis. 2018 Jul;77(7):988-995. doi: 10.1136/annrheumdis-2017-212461. Epub 2018 Feb 20. PMID 29463520
- [Derived] Schiff M, Takeuchi T, Fleischmann R, Gaich CL, DeLozier AM, Schlichting D, Kuo WL, Won JE, Carmack T, Rooney T, Durez P, Shaikh S, Hidalgo RP, van Vollenhoven R, Zerbini CAF. Patient-reported outcomes of baricitinib in patients with rheumatoid arthritis and no or limited prior disease-modifying antirheumatic drug treatment. Arthritis Res Ther. 2017 Sep 18;19(1):208. doi: 10.1186/s13075-017-1410-1. PMID 28923098
- [Derived] Fleischmann R, Schiff M, van der Heijde D, Ramos-Remus C, Spindler A, Stanislav M, Zerbini CA, Gurbuz S, Dickson C, de Bono S, Schlichting D, Beattie S, Kuo WL, Rooney T, Macias W, Takeuchi T. Baricitinib, Methotrexate, or Combination in Patients With Rheumatoid Arthritis and No or Limited Prior Disease-Modifying Antirheumatic Drug Treatment. Arthritis Rheumatol. 2017 Mar;69(3):506-517. doi: 10.1002/art.39953. PMID 27723271

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not respond (nonresponders) to study drug were eligible for rescue treatment beginning at Week 24.
  Nonresponders were defined as lack of improvement of at least 20% in both tender joint count and swollen joint count.
Groups:
- Methotrexate: Methotrexate (MTX) administered orally once weekly with dose ranging from 10 to 20 milligram (mg) per week through Week 52. Participants also received baricitinib placebo orally once daily. Starting at Week 24, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily and MTX orally once weekly.
- Baricitinib + MTX: Baricitinib 4 mg administered orally once daily through Week 52. Participants received MTX orally once weekly with dose ranging from 10 to 20 mg per week through Week 52. Starting at Week 24, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily and MTX orally once weekly.
Period: Treatment Period
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Started | 213 | 160 | 215
Received at Least One Dose of Study Drug | 210 | 159 | 215
Rescued | 26 | 7 | 6
Completed | 161 | 136 | 173
Not Completed | 52 | 24 | 42
Not completed — Withdrawal by Subject | 18 | 7 | 13
Not completed — Lack of Efficacy | 13 | 2 | 2
Not completed — Adverse Event | 8 | 10 | 24
Not completed — Physician Decision | 4 | 3 | 2
Not completed — Death | 3 | 0 | 0
Not completed — Entry Criteria Not Met | 1 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Randomized, Not Treated | 3 | 1 | 0
Period: Follow Up
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Started | 25 (Participants from treatment who entered the post-treatment follow-up period.) | 15 (Participants from treatment who entered the post-treatment follow-up period.) | 28 (Participants from treatment and rescue who entered the post-treatment follow-up period.)
Completed | 0 | 0 | 0
Not Completed | 25 | 15 | 28

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX | Total
Number analyzed (Participants) | 210 | 159 | 215 | 584
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (13.4) | 50.9 (13.0) | 48.5 (13.5) | 49.9 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 121 | 156 | 425
  Male | 62 | 38 | 59 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 10 | 20 | 41
  Asian | 60 | 44 | 61 | 165
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 5 | 10 | 25
  White | 128 | 98 | 123 | 349
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 41 | 29 | 33 | 103
  Austria | 1 | 1 | 1 | 3
  Belgium | 6 | 10 | 11 | 27
  Brazil | 8 | 3 | 9 | 20
  Canada | 5 | 5 | 7 | 17
  Germany | 5 | 5 | 4 | 14
  Greece | 0 | 0 | 1 | 1
  India | 18 | 12 | 17 | 47
  Italy | 8 | 2 | 4 | 14
  Japan | 36 | 29 | 39 | 104
  Mexico | 12 | 14 | 20 | 46
  Portugal | 1 | 0 | 2 | 3
  Russian Federation | 11 | 13 | 12 | 36
  South Africa | 7 | 4 | 9 | 20
  Korea, Republic of | 4 | 1 | 2 | 7
  Sweden | 3 | 0 | 1 | 4
  United Kingdom | 7 | 3 | 4 | 14
  United States | 37 | 28 | 39 | 104
Duration of Rheumatoid Arthritis [Median (Inter-Quartile Range); unit: years] | 0.2 [0.1 to 0.6] | 0.2 [0.1 to 1.1] | 0.2 [0.1 to 1.0] | 0.2 [0.1 to 0.8]
Tender Joint Count of 68 evaluable joints [Mean (Standard Deviation); unit: number of joints] | 26.5 (14.8) | 26.4 (14.1) | 27.7 (14.5) | 26.9 (14.5)
Swollen Joint Count of 66 evaluable joints [Mean (Standard Deviation); unit: number of joints] | 16.4 (10.6) | 16.1 (9.2) | 16.3 (9.5) | 16.3 (9.8)
High sensitivity C-reactive protein [Mean (Standard Deviation); unit: milligrams per liter (mg/L)] | 22.34 (21.78) | 23.75 (26.24) | 24.27 (29.42) | 23.44 (25.98)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Improvement (ACR20)
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). "ACR20 Responder" is a participant who has at least 20% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity using visual analog scale (VAS), Health Assessment Questionnaire-Disability Index (HAQ-DI), pain due to arthritis, and high-sensitivity C-reactive protein (hsCRP). Participants with missing responses and participants who discontinued study or drug or were rescued before analysis time point were deemed non-responders.
Time Frame: Week 24
Population: Modified Intent-to-Treat (mITT) population: all randomized participants who received at least 1 dose of study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using nonresponder imputation (NRI).
Measure: Number; unit: Percent of participants
Groups:
- Methotrexate: MTX administered orally once weekly with dose ranging from 10 to 20 mg per week through Week 52. Participants also received baricitinib placebo orally once daily. Starting at Week 24, participants who were nonresponders were rescued with baricitinib 4 mg orally once daily and MTX orally once weekly.
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
Percent of participants | 61.9 | 76.7 | 78.1
Statistical Analysis 1: Comparison: Methotrexate vs Baricitinib; Test type: Non-Inferiority or Equivalence — Noninferiority is concluded if the lower bound of the 95% CI for the difference in response rate is >-12%; Newcombe-Wilson method = 14.8, 95% CI 2-sided [5.5 to 24.1] — Estimation Parameter: Newcombe-Wilson method without continuity correction for difference in the response rate (Baricitinib minus Methotrexate)

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Improvement (ACR20)
Description: as for outcome 1
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
Percent of participants | 55.7 | 73.0 | 72.6

3. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area are averaged to calculate the HAQ-DI score, which ranges from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicates an improvement in the participant's condition.
Time Frame: Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified baseline observation carried forward (mBOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
units on a scale | -0.73 (0.71) | -1.01 (0.74) | -0.92 (0.74)

4. Secondary Outcome: Change From Baseline in the Disease Activity Score Based on a 28-Joint Count and High-sensitivity C-reactive Protein (DAS28-hsCRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), C-reactive protein (CRP) (milligrams per liter), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using the following formula: DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*Patient's Global VAS+0.96. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mBOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
units on a scale | -2.01 (1.51) | -2.74 (1.39) | -2.82 (1.58)

5. Secondary Outcome: Change From Baseline in the Modified Total Sharp Score (mTSS)
Description: X-rays of the hands/wrists and feet were scored for structural progression as measured using the mTSS (van der Heijde 2000). This methodology quantified the extent of bone erosions and joint space narrowing for 44 and 42 joints, with higher scores representing greater damage.
  The mTSS at a time point is the sum of the erosion (range from 0 to 280) and JSN (range from 0 to 168) scores, for a maximum score of 448.
Time Frame: Baseline, Week 24
Population: mITT population: all randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline assessments. Missing values due to discontinuation of study, rescue, or missing data were imputed using linear extrapolation (LE).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 191 | 152 | 198
units on a scale | 0.64 (1.81) | 0.43 (1.18) | 0.32 (1.14)

6. Secondary Outcome: Percentage of Participants Who Achieved a Simplified Disease Activity Index (SDAI) Score ≤3.3
Description: SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Patient's Global Assessment of Disease Activity using VAS centimeters (cm), and Physician's Global Assessment of Disease Activity using VAS (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity. An index-based definition of remission occurs with an SDAI score ≤3.3.
Time Frame: Week 24
Population: mITT population: all randomized participants who received at least 1 dose of study drug. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using NRI.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
percentage of participants | 10.5 | 22.0 | 22.8

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 Responder Index is composite of clinical, laboratory, and functional measures in RA. "ACR50 Responder" is a participant who has at least 50% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinued study or drug or were rescued before analysis time point were deemed non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: as for outcome 6
Measure: Number; unit: Percent of participants
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
Percent of participants
  Week 12 | 32.9 | 54.7 | 60.0
  Week 24 | 43.3 | 59.7 | 63.3
  Week 52 | 37.6 | 57.2 | 61.9

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 Responder Index is composite of clinical, laboratory, and functional measures in RA. "ACR70 Responder" is a participant who has at least 70% improvement in both tender and swollen joint counts and in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, HAQ-DI, pain due to arthritis, and hsCRP. Participants with missing responses and participants who discontinued study or drug or were rescued before analysis timepoint were deemed non-responders.
Time Frame: Week 12, Week 24, Week 52
Population: as for outcome 6
Measure: Number; unit: Percent of participants
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
Percent of participants
  Week 12 | 15.7 | 30.8 | 33.5
  Week 24 | 21.4 | 42.1 | 39.5
  Week 52 | 25.2 | 42.1 | 46.0

9. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score
Description: The CDAI is a tool for measurement of disease activity in RA that does not require a laboratory component and was scored by the investigative site. It integrates TJC28 (scored 0-28 with higher scores indicating higher disease activity), SJC28 (scored 0-28 with higher scores indicating higher disease activity), Patient's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity), and Physician's Global Assessment of Disease Activity (scored on a visual analogue scale from 0-10 cm with higher scores indicating higher disease activity). The CDAI is calculated by summing the values of the 4 components. CDAI scores range from 0 to 76; lower scores indicated lower disease activity. A negative change from baseline indicates improvement in condition.
Time Frame: Baseline, Week 24; Baseline, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using modified last observation carried forward (mLOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 200 | 157 | 208
units on a scale
  Week 24 | -22.12 (16.12) | -28.20 (13.96) | -29.86 (14.05)
  Week 52 | -21.95 (18.07) | -28.94 (14.58) | -30.72 (14.87)

10. Secondary Outcome: Change From Baseline in Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: DAS28 consisted of a composite score of the following variables: tender joint count (TJC28), swollen joint count (SJC28), erythrocyte sedimentation rate (ESR) (millimeters per hour), and Patient's Global Assessment of Disease Activity. DAS28 was calculated using the following formula: DAS28-ESR=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.70*natural log(ESR)+0.014*Patient's Global VAS. Scores ranged 1.0-9.4, where lower scores indicated less disease activity.
Time Frame: Baseline, Week 24; Baseline, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug, with a baseline value and at least 1 post-baseline value. Missing values due to discontinuation of study or drug, rescue, or missing data were imputed using mLOCF.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 203 | 159 | 209
units on a scale
  Week 24 | -2.20 (1.53) | -2.76 (1.45) | -3.06 (1.46)
  Week 52 | -2.32 (1.77) | -2.84 (1.57) | -3.22 (1.48)

11. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Remission
Description: The ACR/EULAR definitions of RA remission include a "Boolean-based definition". The Boolean-based definition of remission occurs when all 4 of the following criteria are met at the same visit: TJC28 ≤1, SJC28 ≤1, acute phase response using C-reactive protein (milligrams per deciliter) ≤1, Patient's Global Assessment of Disease Activity using VAS (cm) ≤1.
Time Frame: Week 12, Week 24, Week 52
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
percentage of participants
  Week 12 | 5.7 | 13.8 | 14.4
  Week 24 | 8.6 | 18.9 | 16.3
  Week 52 | 11.4 | 17.0 | 20.9

12. Secondary Outcome: Change From Baseline in Joint Space Narrowing and Bone Erosion Scores
Description: X-rays of the hands/wrists and feet were assessed for joint space narrowing (JSN) and bone erosions. Assessment of JSN for each hand (15 joints per hand) and foot (6 joints per foot), including subluxation, is scored from 0 to 4, with 0 indicating no (normal) JSN and 4 indicating complete loss of joint space, bony ankylosis or luxation. JSN scores ranged from 0-168. A score of 0 would indicate no change and higher scores represent a worsening of joint space narrowing. The bone erosion score is a summary of erosion severity in 32 joints of the hands and 12 joints of the feet. Each joint is scored according to the surface area involved from 0 to 5 for hand joints and 0 to 10 for the foot joints, with 0 indicating no erosion and the highest score (5 for the hand and 10 for the foot) indicating extensive loss of bone from more than one half of the articulating bone. Erosion scores ranged from 0 (no erosion) to 280 (high erosion).
Time Frame: Baseline, Week 24; Baseline, Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-baseline assessment. Missing values due to discontinuation of study, rescue, or missing data were imputed using LE.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
units on a scale
  JSN Week 24: number analyzed (Participants) | 191 | 152 | 198
  JSN Week 24 | 0.15 (0.94) | 0.08 (0.44) | 0.05 (0.44)
  JSN Week 52: number analyzed (Participants) | 192 | 154 | 199
  JSN Week 52 | 0.23 (1.00) | 0.26 (1.14) | 0.08 (0.88)
  Bone Erosion Week 24: number analyzed (Participants) | 191 | 152 | 198
  Bone Erosion Week 24 | 0.49 (1.14) | 0.35 (0.92) | 0.27 (0.95)
  Bone Erosion Week 52: number analyzed (Participants) | 192 | 154 | 199
  Bone Erosion Week 52 | 0.80 (1.80) | 0.55 (1.48) | 0.33 (1.21)

13. Secondary Outcome: Change From Baseline in Duration of Morning Joint Stiffness
Description: Participants reported the duration of their morning joint stiffness (MJS) in hours and minutes. The participants were asked about their duration of morning joint stiffness on the day prior to the study visit to capture actual symptoms, since the participant may have had an atypical morning routine on the day of the study visit. If morning joint stiffness duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. A decrease in duration of morning joint stiffness indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 52
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 204 | 159 | 209
Minutes | -40.0 [-55.0 to -30.0] | -55.0 [-60.0 to -40.0] | -60.0 [-80.0 to -50.0]

14. Secondary Outcome: Change From Baseline in Worst Tiredness Numeric Rating Scale (NRS)
Description: Participants rated their tiredness by selecting a number from 0 to 10 that best described their worst tiredness during the last 24 hours, where 0 represents "no tiredness" and 10 represents "as bad as you can imagine".
Time Frame: Baseline, Week 24; Baseline Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 204 | 159 | 209
units on a scale
  Week 24 | -2.2 (2.7) | -3.0 (3.1) | -3.0 (2.8)
  Week 52 | -2.3 (2.8) | -2.9 (3.1) | -3.0 (2.9)

15. Secondary Outcome: Change From Baseline in Worst Joint Pain Numeric Rating Scale (NRS)
Description: Participants rated their joint pain by selecting a number from 0 to 10 that best described their worst joint pain during the last 24 hours, where 0 represents "no pain" and 10 represents "pain as bad as you can imagine".
Time Frame: Baseline, Week 24; Baseline Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 204 | 159 | 209
units on a scale
  Week 24 | -2.8 (2.5) | -3.9 (2.7) | -3.9 (2.6)
  Week 52 | -3.0 (2.8) | -3.9 (2.9) | -4.1 (2.7)

16. Secondary Outcome: Change From Baseline in Mental Component Score (MCS) and Physical Component Score (PCS) of the Medical Outcomes Study 36-Item Short Form Health Survey Version 2 Acute (SF-36v2 Acute)
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains: physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, and 2 component scores (MCS and PCS). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with higher scores indicating better health status or functioning.
Time Frame: Baseline, Week 24; Baseline Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 202 | 159 | 207
units on a scale
  MCS Week 24 | 3.4 (10.8) | 5.9 (11.7) | 4.6 (11.6)
  MCS Week 52 | 2.4 (10.9) | 5.8 (11.9) | 5.0 (11.5)
  PCS Week 24 | 9.4 (9.2) | 12.5 (9.1) | 13.2 (9.6)
  PCS Week 52 | 9.4 (10.1) | 11.6 (9.6) | 13.3 (9.8)

17. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores
Description: European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a standardized measure of health status of the participant. One component consists of a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state.
Time Frame: Baseline, Week 24; Baseline Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 202 | 159 | 207
units on a scale
  Index Score (US Algorithm) Week 24 | 0.142 (0.189) | 0.197 (0.164) | 0.194 (0.180)
  Index Score (US Algorithm) Week 52 | 0.138 (0.203) | 0.186 (0.177) | 0.185 (0.186)
  Index Score (UK Algorithm) Week 24 | 0.205 (0.274) | 0.285 (0.241) | 0.282 (0.255)
  Index Score (UK Algorithm) Week 52 | 0.197 (0.294) | 0.271 (0.258) | 0.268 (0.266)

18. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) Scores (Self-Perceived Health)
Description: A second component of the EQ-5D-5L is a self-perceived health score which is assessed using a VAS that ranges from 0 to 100 millimeter (mm), where 0 indicates the worst health you can imagine and 100 indicates the best health you can imagine.
Time Frame: Baseline, Week 24; Baseline Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 202 | 159 | 207
millimeter
  Self-Perceived Health Week 24 | 14.5 (28.3) | 24.1 (26.0) | 21.4 (31.4)
  Self-Perceived Health Week 52 | 13.6 (30.1) | 24.5 (28.7) | 24.5 (30.6)

19. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scores
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale is a13-item, symptom-specific questionnaire that specifically assesses the participant's self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses a numeric rating scale of 0 ("Not at all") to 4 ("Very much") for each item to assess fatigue and its impact in the past 7 days. Total scores range from 0 to 52, with higher scores indicating less fatigue.
Time Frame: Baseline, Week 24; Baseline Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 204 | 159 | 209
units on a scale
  Week 24 | 9.3 (11.2) | 13.0 (10.8) | 12.3 (11.5)
  Week 52 | 9.1 (10.9) | 11.3 (10.8) | 12.6 (11.8)

20. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) Scores
Description: The Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA) questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. It contains 6 items covering overall work productivity (health), overall work productivity (symptom), impairment of regular activities (health), and impairment of regular activities (symptom). Scores are calculated as impairment percentages. The WPAI-RA yields four types of scores: Absenteeism (work time missed), Presenteeism (impairment at work), Work productivity loss (overall work impairment), and Activity impairment.
Time Frame: Baseline, Week 24; Baseline Week 52
Population: mITT population: all randomized participants who received at least 1 dose of study drug, with a baseline value and an observed value at the time point being summarized.
Measure: Mean (Standard Deviation); unit: Percentage of Impairment
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX
Number analyzed (Participants) | 210 | 159 | 215
Percentage of Impairment
  Absenteeism Week 24 (n=76, 56, 90) | -3.6 (35.5) | -8.7 (30.4) | -7.6 (26.5)
  Absenteeism Week 52 (n=52, 51, 71) | -3.0 (29.2) | -8.4 (29.7) | -7.3 (21.8)
  Presenteeism Week 24(n=70, 51, 86) | -19 (25) | -26 (27) | -32 (26)
  Presenteeism Week 52 (n=51, 47, 75) | -26 (26) | -27 (24) | -33 (25)
  Work Productivity Loss Week 24 (n=70, 71, 86) | -17.8 (30.2) | -25.6 (29.1) | -30.9 (29.6)
  Work Productivity Loss Week 52 (n=51, 47, 75) | -24.1 (30.5) | -27.6 (27.3) | -33.8 (27.5)
  Activity Impairment Week 24 (n=184, 145, 192) | -25 (26) | -36 (28) | -31 (28)
  Activity Impairment Week 52 (n=141, 131, 172) | -28 (27) | -34 (27) | -37 (27)

21. Secondary Outcome: Population Pharmacokinetics (PK): Peak Concentration at Steady State (Cmax,ss) of Baricitinib
Time Frame: Week 0: 15 and 60 minutes postdose; Week 4: 2 to 4 hours post-dose; Week 8: 4 to 6 hours post-dose; Week 12; Week 24; Week 32; Pre-dose
Population: All randomized participants who received at least 1 dose of study drug (during study or rescue treatment) with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | Baricitinib
Number analyzed (Participants) | 355
nanomole/Liter (nmol/L) | 135 (23.1)

22. Secondary Outcome: Population PK: Area Under the Concentration Versus Time Curve at a Dosing Interval at Steady State (AUCtau,ss) of Baricitinib
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | Baricitinib
Number analyzed (Participants) | 355
nanomole/Liter (nmol/L) | 1280 (47.2)

ADVERSE EVENTS:
Description: All enrolled participants including those receiving rescue therapy, with events occurring after rescue accounted separately. Rescue therapy occurred at Week 24 or later, if determined to be nonresponders (lack of improvement of at least 20% in both tender joint count and swollen joint count).
Groups:
- Rescue Period: Baricitinib 4 mg administered orally once daily through Week 52. Participants received MTX orally once weekly with dose ranging from 10 to 20 mg per week through Week 52.
- Methotrexate - Follow-up; Baricitinib - Follow-up: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug.
- Baricitinib + MTX - Follow-up: No study drug received. Participants return for safety follow-up visit 28 days after the last dose of study drug. Includes participants who were rescued to Baricitinib + MTX.
Arm/Group | Methotrexate | Baricitinib | Baricitinib + MTX | Rescue Period | Methotrexate - Follow-up | Baricitinib - Follow-up | Baricitinib + MTX - Follow-up
Serious Adverse Events (participants affected / at risk) | 20/210 | 12/159 | 17/215 | 1/39 | 0/25 | 0/15 | 0/28
Other Adverse Events (participants affected / at risk) | 115/210 | 81/159 | 129/215 | 21/39 | 2/25 | 2/15 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=210) | Baricitinib (N=159) | Baricitinib + MTX (N=215) | Rescue Period (N=39) | Methotrexate - Follow-up (N=25) | Baricitinib - Follow-up (N=15) | Baricitinib + MTX - Follow-up (N=28)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder adenosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Methotrexate (N=210) | Baricitinib (N=159) | Baricitinib + MTX (N=215) | Rescue Period (N=39) | Methotrexate - Follow-up (N=25) | Baricitinib - Follow-up (N=15) | Baricitinib + MTX - Follow-up (N=28)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3) | 7 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scleromalacia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (20) | 16 (21) | 21 (32) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (6) | 2 (2) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 12 (14) | 16 (19) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1/28 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1) | 13 (15) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 4 (5) | 10 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 9 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1/28 (1) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 5 (7) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 2 (2) | 13 (13) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (16) | 7 (7) | 20 (26) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 5 (5) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (5) | 3 (3) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 5 (5) | 1 (1) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 5 (5) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 10 (10) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 7 (7) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 7 (7) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 5 (5) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 6 (7) | 14 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/148 (1) | 0 (0) | 6/156 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (6) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days